CLINICAL TRIAL: NCT00160368
Title: Effect of Potassium Bicarbonate and Potassium Chloride on Blood Pressure and Markers of Target Organ Damage in Hypertensives
Brief Title: Effects of Potassium Salts on Blood Pressure and Target Organ Damage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CH/FR/04.0012
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Hypertension
Keywords: Hypertension, potassium salts
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Potassium supplementation

SUMMARY:
The purpose of this study is to determine the effect of potassium chloride and potassium bicarbonate on blood pressure and also to determine whether increasing potassium intake has beneficial effects on the surrogate markers of target organ damage in cardiovascular disease, as well as on bone health.

DETAILED DESCRIPTION:
Randomised trials have shown that increasing potassium intake lowers blood pressure. However, most previous trials used potassium chloride. Whereas, potassium in fruits and vegetables is not a chloride salt, but a mixture of potassium phosphate, sulphate, citrate, and many organic anions, most of which are precursors of potassium bicarbonate. It is unclear whether non-chloride salt of potassium has greater or lesser effect on blood pressure compared to potassium chloride.

Experimental studies in animals and epidemiological studies in humans suggest that a high potassium intake may have beneficial effects on the cardiovascular system and the kidney, independent of its effect on blood pressure, and also reduce the risk of osteoporosis.

We propose to carry out a randomised double-blind trial to compare potassium bicarbonate with potassium chloride looking at their effect on blood pressure, and also to determine whether these potassium salts have beneficial effects on the cardiovascular system, kidney and bone health.

Comparisons: potassium chloride vs potassium bicarbonate vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated essential hypertension (sitting systolic blood pressure between 140 and 170 mmHg and/or sitting diastolic blood pressure between 90 and 105 mmHg);
* Age 18 - 75 years.

Exclusion Criteria:

* Individuals younger than 18 or older than 75 years;
* Individuals with impaired renal function with plasma creatinine greater than 120 umol/L for non-blacks or 150 umol/L for blacks;
* Individuals with chronic diarrhea, or history of peptic ulcer;
* Individuals with baseline plasma potassium values greater than 5.0 mmol/L;
* Individuals with severe hypertension i.e. blood pressure > 170/105 mmHg;
* Individuals with diabetes mellitus;
* Individuals with any secondary cause of hypertension;
* Individuals with malignancy or liver disease;
* Individuals with ischaemic heart disease or heart failure;
* Females who are pregnant or breast feeding or on the oral contraceptive pill.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-01; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure and markers of target organ damage and bone health at 4 weeks of potassium supplementation.

SECONDARY OUTCOMES:
Comparisons among different treatments in blood pressure and markers of target organ damage and bone health.

CONTACTS AND LOCATIONS:
Overall Officials: Graham A MacGregor, MD, Principal Investigator — St George's, University of London
Locations (1):
- St. George's University of London,, London, United Kingdom